CLINICAL TRIAL: NCT02138500
Title: A Phase 1, Open-label Study To Evaluate Central Occupancy Of The Benzodiazepine Binding Site Of Gabaa Receptors By Positron Emission Tomography (Pet) With Ligand [11c]Flumazenil Following Single Dose Of Pf-06372865 In Healthy Subjects
Brief Title: A Study to Examine the Distribution of PF-06372865 in the Brain of Healthy Volunteers Using Positron Emission Tomography and a Radioactive Tracer Following Oral Administration of One Dose of PF-06372865
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B7431004
Record Dates: First submitted 2014-04-08; First posted 2014-05-14 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
Keywords: PF-06372865; phase 1; open-label; GABA-A receptor occupancy; positron emission tomography; healthy subjects
MeSH Terms: interventions — PF-06372865

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1: PF-06372865 10 mg (Experimental)
  Interventions: Drug: PF-06372865
- Cohort 2: PF-06372865 TBD dose (Experimental)
  Interventions: Drug: PF-06372865
- Cohort 3: PF-06372865 TBD dose (Experimental)
  Interventions: Drug: PF-06372865

INTERVENTIONS:
Drug: PF-06372865 — Single, oral dose administration of 10 mg PF-06372865 using tablet formulation.
  Arms: Cohort 1: PF-06372865 10 mg
Drug: PF-06372865 — Single, oral dose administration of TBD dose PF-06372865 using tablet/extemprep formulation.
  Arms: Cohort 2: PF-06372865 TBD dose
Drug: PF-06372865 — Single, oral dose administration of TBD dose PF-06372865 using tablet/extemprep formulation.
  Arms: Cohort 3: PF-06372865 TBD dose

SUMMARY:
This study will see how PF-06372865, an experimental drug distributes in the brain after one dose of PF-06372865 is administered orally to healthy volunteer subjects. The study will also evaluate the safety and tolerability of PF-06372865in these subjects and will measure the level of PF-06372865 in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects and female subjects of non-childbearing potential between the ages of 18 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* Known or suspected sensitivity to flumazenil and other benzodiazepines.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
GABAA RO in the whole brain | Change from baseline to days 1 and 2
Average plasma concentration of PF-06372865 in post-dose PET scans after single oral doses of PF-06372865 | Change from baseline to days 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - New Haven Clinical Research Unit, New Haven, Connecticut
  - Anlyan Center, New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7431004&StudyName=A%20Study%20to%20Examine%20the%20Distribution%20of%20PF-06372865%20in%20the%20Brain%20of%20Healthy%20Volunteers%20Using%20Positron%20Emission%20Tomography%20and%20a%20Radioac